CLINICAL TRIAL: NCT07170267
Title: Analgesic Efficacy of Transversalis Fascia Plane Block Versus Intrathecal Dexmedetomidine in Patients Undergoing Cesarean Section: A Randomized Controlled Trial
Brief Title: Transversalis Fascia Plane Block Versus Intrathecal Dexmedetomidine in Patients Undergoing Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1335/8/25
Record Dates: First submitted 2025-09-06; First posted 2025-09-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Transversalis Fascia Plane Block; Intrathecal Dexmedetomidine; Cesarean Section

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TFP group (Experimental): Patients will receive spinal anesthesia (using 2.5 mL of hyperbaric bupivacaine 0.5%) with bilateral transversalis fascia plane (TFP) block (using 20 mL of bupivacaine 0.25%) at the end of surgery.
  Interventions: Other: Transversalis fascia plane block
- Control group (Active Comparator): Patients will receive spinal anesthesia (using 2.5 mL of hyperbaric bupivacaine 0.5%) + (5 µg intrathecal dexmedetomidine diluted in 0.5ml saline) with a sham block at the end of surgery.
  Interventions: Drug: Intrathecal dexmedetomidine

INTERVENTIONS:
Other: Transversalis fascia plane block — Patients will receive spinal anesthesia (using 2.5 mL of hyperbaric bupivacaine 0.5%) with bilateral transversalis fascia plane (TFP) block (using 20 mL of bupivacaine 0.25%) at the end of surgery.
  Arms: TFP group
Drug: Intrathecal dexmedetomidine — Patients will receive spinal anesthesia (using 2.5 mL of hyperbaric bupivacaine 0.5%) + (5 µg intrathecal dexmedetomidine diluted in 0.5ml saline) with a sham block at the end of surgery.
  Arms: Control group

SUMMARY:
This study aims to compare the analgesic efficacy of the transversalis fascia plane (TFP) block and intrathecal dexmedetomidine in patients undergoing cesarean section (CS).

DETAILED DESCRIPTION:
Cesarean section (CS) is a commonly performed major surgical procedure that results in substantial postoperative pain and patient dissatisfaction.

Spinal anesthesia is commonly used in CS surgery. However, it may be associated with several side effects, particularly hypotension.

Dexmedetomidine is an α2 adrenergic receptor agonist that has an analgesic effect.

Ultrasound-guided interfascial plane blocks are often used in multimodal analgesia regimens. Local anaesthetic injection into the transversalis fascia plane (TFP) anesthetizes the proximal branches of T12 and L1 which targeted in the plane between the transversus abdominis muscle and the transversalis fascia.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 40 years.
* American Society of Anesthesiology (ASA) physical status II.
* Women undergoing cesarean section under spinal anesthesia.

Exclusion Criteria:

* Contraindication to spinal anesthesia.
* Women with body mass index >40 kg/m2.
* Pregnancy-induced hypertension
* Local infection at the site of injection.
* Known cardiovascular disease
* Coagulation abnormality.
* History of chronic pain.
* Abuse of drugs or alcohol.
* History of allergies to any study medications.
* Seizure disorders.
* Any pregnancy complications requiring conversion to general anesthesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing cesarean section
Enrollment: 50 (Estimated)
Dates: Start 2025-09-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at post-anesthesia care unit (PACU), 2, 4, 6, 8, 12, 18 and 24 h postoperatively.

SECONDARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4.
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia will be recorded from the end of surgery to first dose of morphine administrated.
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded preoperatively and every 30 minutes till the end of surgery.
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded preoperatively and every 30 minutes till the end of surgery.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.